CLINICAL TRIAL: NCT03988985
Title: Enhancing the Clinical Effectiveness of Depression Screening Using Patient-targeted Feedback in General Practices: The GET.FEEDBACK.GP Multicentre Randomized Controlled Trial
Brief Title: Enhancing the Clinical Effectiveness of Depression Screening Using Patient-targeted Feedback in General Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Federal Joint Committee (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: UHHamburgEppendorfGetFeedback
Record Dates: First submitted 2019-06-04; First posted 2019-06-18 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Depression
Keywords: Depression; Screening; Primary Care; General Practice; Feedback
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PATIENT-GP-FEEDBACK (Experimental): Using a randomized-controlled study design one third of the patients and their attending general practitioner will receive feedback after depression screening. The feedback for the patient contains the screening result, information about depression in general, guideline based treatment recommendations for patients and contact-information for treatment. The feedback for the general practitioner contains the screening result and guideline-based recommendations, i.e. to inform patients of their depression screening result. Nevertheless, in order to reflect routine clinical practice, the physicians will decide themselves whether or not to address depression during their consultation with the patient.
  Interventions: Other: Patient-targeted feedback; Other: GP-targeted feedback
- GP-FEEDBACK (Active Comparator): Using a randomized-controlled study design in one third of the cases only the attending general practitioner will receive feedback after depression screening. The feedback for the general practitioner contains the screening result and guideline-based recommendations, i.e. to inform patients of their depression screening result. Nevertheless, in order to reflect routine clinical practice, the physicians will decide themselves whether or not to address depression during their consultation with the patient.
  Interventions: Other: GP-targeted feedback
- NO-FEEDBACK (No Intervention): Using a randomized-controlled study design one third of the patients and their attending general practitioner will not receive any feedback.

INTERVENTIONS:
Other: Patient-targeted feedback — The feedback for the patient contains the screening result, information about depression in general, guideline based treatment recommendations for patients and contact-information for treatment.
  Arms: PATIENT-GP-FEEDBACK
Other: GP-targeted feedback — The feedback for the general practitioner contains the screening result and guideline-based recommendations, i.e. to inform patients of their depression screening result. Nevertheless, in order to reflect routine clinical practice, the physicians will decide themselves whether or not to address depression during their consultation with the patient.
  Arms: GP-FEEDBACK; PATIENT-GP-FEEDBACK

SUMMARY:
The multi-center GET.FEEDBACK.GP randomized controlled trial is designed based on patients' needs and preferences. In order to evaluate the effect of feedback in the broader setting of primary care, a total of 1076 primary care patients with elevated levels of depression (PHQ-9 score ≥ 10) will be randomized into three groups who either receive a) patient-targeted and physician-targeted feedback of depression screening results, b) a physician-targeted feedback of depression screening results only, or c) no feedback of screening results. The primary study outcome is depression severity after 6 months, secondary outcomes include the patients' behavior and cognitions after the screening, depression care according to German guideline recommendations and the health economic evaluation.

DETAILED DESCRIPTION:
Major depression is one of the most significant clinical disorders. In primary care, every sixth patient suffers from increased depression level, which is associated with higher risk of suicide, increased risk of onset and progression of chronic physical conditions. Still, depression is under recognized and undertreated in primary care. Moreover, evidence regarding the efficacy of depression screening in primary care is insufficient to draw clear conclusions. Our previous mono-center depression screening trial in cardiac patients, provides first evidence that written patient-targeted feedback improves depression severity, encourages greater patient participation and engagement in mental health. To amplify these effects, the multi-center GET.FEEDBACK.GP randomized controlled trial is now designed based on patients' needs and preferences. In order to evaluate the effect of feedback in the broader setting of primary care, a total of 1076 primary care patients with elevated levels of depression (PHQ-9 score ≥ 10) will be randomized into three groups who either receive a) patient-targeted and physician-targeted feedback of depression screening results, b) a physician-targeted feedback of depression screening results only, or c) no feedback of screening results. The primary study outcome is depression severity after 6 months, secondary outcomes include the patients' behavior and cognitions after the screening, depression care according to German guideline recommendations and the health economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male, female, diverse
* Maximum Age: no maximum age
* Attendance in primary care with medical consultation
* Age ≥ 18 years;
* Sufficient language skills;
* Informed consent
* Patient Health Questionnaire-9 > 9 points

Exclusion Criteria:

* Life threatening health status;
* Severe somatic or/and psychological disorder that needs urgent treatment;
* Known diagnosis of a depressive disorder
* Current depression treatment
* Acute suicidal tendency;
* Severe cognitive or/and visual difficulties;
* Not being able to fill out questionnaires
* No contact details

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Depression severity (Questionnaire: Patient Health Questionnaire-9) | Six months after screening
  Level of depression severity six months after screening (Patient Health Questionnaire-9)

SECONDARY OUTCOMES:
Depression severity (Questionnaire: Patient Health Questionnaire-9) | One and twelve months after screening
  Level of depression severity one and twelve months after screening (Questionnaire: Patient Health Questionnaire-9)
Depression treatment | Six and twelve months after screening
  Proportion of patients treated according to German Guideline based recommendations
Health economic Evaluation (Questionnaire: Client Sociodemographic and Service Receipt Inventory) | Six and twelve months after screening
  Direct and indirect health costs (Client Sociodemographic and Service Receipt Inventory)
Quality-adjusted life years (Questionnaire: EuroQol-5D) | Six and twelve months after screening
  Quality-adjusted years of life and quality of life (EuroQol-5D)
Anxiety (Questionnaire: Generalized Anxiety Disorder-7) | One, six and twelve months after screening
  Level of anxiety severity one, six and twelve months after screening
Somatic symptom severity (Questionnaire: Somatic Symptom Scale-8) | One, six and twelve months after screening
  Level of somatic symptom severity one, six and twelve months after screening

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Löwe, MD, Principal Investigator — Director of the Department of Psychosomatic Medicine and Psychotherapy
Locations (5):
- Germany (5):
  - University Medical Center Heidelberg, Heidelberg, Baden-Würtenberg
  - University Medical Center Tuebingen, Tübingen, Baden-Würtenberg
  - Technical University of Munich - Medical Faculty, Munich, Bavaria
  - University Medical Center Jena, Jena, Thuringia
  - University Medical Center Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the ethics approval of the Ethics Committee of the Hamburg Medical Association on April 8, 2019, (approval number PV6031) and the German Research Foundation guidelines for the handling of research data, deidentified data will be made available on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available six months after publication of the main findings. Data will be available for ten years after publication of the main findings.
Access Criteria: Data can be requested by the principal investigators. Data use and request underly the publication policy of the multicentre GET.FEEBDACK.GP RCT.

REFERENCES:
- [Background] Kohlmann S, Lehmann M, Eisele M, Braunschneider LE, Marx G, Zapf A, Wegscheider K, Harter M, Konig HH, Gallinat J, Joos S, Resmark G, Schneider A, Allwang C, Szecsenyi J, Nikendei C, Schulz S, Brenk-Franz K, Scherer M, Lowe B. Depression screening using patient-targeted feedback in general practices: study protocol of the German multicentre GET.FEEDBACK.GP randomised controlled trial. BMJ Open. 2020 Sep 21;10(9):e035973. doi: 10.1136/bmjopen-2019-035973. PMID 32958483
- [Derived] Kreis LG, Konig HH, Kohlmann S, Lowe B, Scherer M, Brettschneider C. Cost-effectiveness of targeted feedback interventions after depression screening in primary care: health economic evaluation of the GET.FEEDBACK.GP trial. BJPsych Open. 2026 Feb 2;12(2):e52. doi: 10.1192/bjo.2025.10945. PMID 41621811
- [Derived] Lowe B, Scherer M, Braunschneider LE, Marx G, Eisele M, Mallon T, Schneider A, Linde K, Allwang C, Joos S, Zipfel S, Schulz S, Rost L, Brenk-Franz K, Szecsenyi J, Nikendei C, Harter M, Gallinat J, Konig HH, Fierenz A, Vettorazzi E, Zapf A, Lehmann M, Kohlmann S. Clinical effectiveness of patient-targeted feedback following depression screening in general practice (GET.FEEDBACK.GP): an investigator-initiated, prospective, multicentre, three-arm, observer-blinded, randomised controlled trial in Germany. Lancet Psychiatry. 2024 Apr;11(4):262-273. doi: 10.1016/S2215-0366(24)00035-X. Epub 2024 Feb 29. PMID 38432236

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03988985/SAP_000.pdf